CLINICAL TRIAL: NCT02085135
Title: A Phase 3, Randomized, Double-blind Study to Evaluate the Safety and Tolerability of Two Titration Schedules for ALKS 5461 for the Adjunctive Treatment of Major Depressive Disorder in Adults With an Inadequate Response to Antidepressant Therapy (the FORWARD-1 Study)
Brief Title: A Study of Different Titration Schedules of ALKS 5461 in Adults With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK5461-210
Record Dates: First submitted 2014-03-07; First posted 2014-03-12 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder
Keywords: depression; major depressive disorder; Alkermes; ALKS 5461; samidorphan; buprenorphine
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — ALKS 5461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Titration Schedule 1 (Experimental)
  Interventions: Drug: ALKS 5461
- Titration Schedule 2 (Experimental)
  Interventions: Drug: ALKS 5461

INTERVENTIONS:
Drug: ALKS 5461 — Sublingual tablet taken once daily

SUMMARY:
This is a Phase 3 study designed to evaluate the safety and tolerability of two titration schedules for ALKS 5461.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18-40 kg/m2
* Have a diagnosis of MDD
* Have a current major depressive episode (MDE) lasting 8 weeks to 24 months
* Have been treated with an adequate dose of an approved antidepressant during the current MDE for at least 8 weeks
* Have an inadequate response to current antidepressant treatment
* Agree to use an approved method of birth control for the duration of the study
* Additional criteria may apply

Exclusion Criteria:

* Currently pregnant or breastfeeding
* History of or current infection with Hepatitis B Virus, Hepatitis C Virus or Human Immunodeficiency Virus (HIV)
* Have experienced hallucinations, delusions, or any psychotic symptoms in the current MDE
* Have used opioid agonists (eg, codeine, oxycodone, tramadol, or morphine) or opioid antagonists (eg, naloxone, naltrexone) within 14 days
* Have received electroconvulsive therapy treatment within the last 5 years
* Have attempted suicide within the past 2 years
* Have a history of intolerance, allergy, or hypersensitivity to buprenorphine or opioid antagonists (eg, naltrexone, naloxone)
* Have had a significant blood loss or blood donation with 60 days of screening
* Additional criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Pathak, MD, Study Director — Alkermes, Inc.
Locations (9):
- United States (8):
  - Alkermes Investigational Site, Jacksonville, Florida
  - Alkermes Investigational Site, Orlando, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Saint Charles, Missouri
  - Alkermes Investigational Site, Staten Island, New York
  - Alkermes Investigational Site, Dayton, Ohio
  - Alkermes Investigational Site, Allentown, Pennsylvania
  - Alkermes Investigational Site, Bellevue, Washington
- Alkermes Investigational Site, Halifax, Nova Scotia, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were diagnosed with major depressive disorder (MDD) and had an inadequate response to 1 or 2 adequate courses of treatment with a commercially available antidepressant therapy (ADT) during the current major depressive episode (MDE). All subjects continued ADT for the duration of the study.
Groups:
- 1-Week Titration: ALKS 5461: Sublingual tablet taken once daily in ascending doses over a 1-week titration period
- 2-Week Titration: ALKS 5461: Sublingual tablet taken once daily in ascending doses over a 2-week titration period
Period: Overall Study
Arm/Group | 1-Week Titration | 2-Week Titration
Started | 34 | 32
Completed | 23 | 23
Not Completed | 11 | 9
Not completed — Adverse Event | 4 | 7
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lack of Efficacy | 2 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-Week Titration | 2-Week Titration | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (12.6) | 50.8 (11.3) | 49.7 (53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 14 | 11 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 32 | 27 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 6 | 14
  White | 24 | 23 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1 | 0 | 1
  United States | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs)
Time Frame: 8 weeks
Population: Number of subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1-Week Titration | 2-Week Titration
Number analyzed (Participants) | 34 | 32
Participants | 27 | 28

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Arm/Group | 1-Week Titration | 2-Week Titration
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32
Other Adverse Events (participants affected / at risk) | 23/34 | 28/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-Week Titration (N=34) | 2-Week Titration (N=32)
Constipation (Gastrointestinal disorders) | 6 (6) | 11 (12)
Nausea (Gastrointestinal disorders) | 9 (14) | 7 (7)
Dry Mouth (Gastrointestinal disorders) | 3 (3) | 8 (8)
Vomiting (Gastrointestinal disorders) | 7 (7) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (12) | 4 (4)
Somnolence (Nervous system disorders) | 3 (3) | 5 (7)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 4 (4) | 1 (1)
Sedation (Nervous system disorders) | 0 (0) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4) | 4 (4)
Fatigue (General disorders) | 6 (6) | 1 (1)
Irritability (General disorders) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Influenza (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.